CLINICAL TRIAL: NCT06670300
Title: Clinical Observation on the Safety and Efficacy of Cardonilmab in the Treatment of Second-line and Above Advanced Melanoma and Advanced Renal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: YongZhang (Other Government)
Responsible Party: Sponsor-Investigator, YongZhang, Immunotherapy Department, Henan Cancer Hospital
Organization: Henan Cancer Hospital (Other Government)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-011
Record Dates: First submitted 2024-10-10; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Participants Who Had Received Second-line or Higher Advanced Melanoma and Advanced Renal Cancer
Keywords: melanoma; renal cancer; Cardonilizumab
MeSH Terms: conditions — Melanoma; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Melanoma and kidney cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cardonilimab for advanced melanoma (Experimental): Subjects will receive cardonilimab 10mg/kg once every three weeks; The maximum duration of administration is 2 years until disease progression or death, toxicity becomes intolerable, subject voluntarily requests withdrawal, or investigator determines that subject needs to withdraw from the study.
  Interventions: Drug: cardonilimab
- cardonilimab for advanced kidney cancer (Experimental): Subjects will receive cardonilimab 10mg/kg once every three weeks; The maximum duration of administration is 2 years until disease progression or death, toxicity becomes intolerable, subject voluntarily requests withdrawal, or investigator determines that subject needs to withdraw from the study.
  Interventions: Drug: cardonilimab

INTERVENTIONS:
Drug: cardonilimab — Subjects will receive cardonilimab 10mg/kg once every three weeks; The maximum duration of administration is 2 years until disease progression or death, toxicity becomes intolerable, subject voluntarily requests withdrawal, or investigator determines that subject needs to withdraw from the study.

SUMMARY:
Safety and efficacy of Cardonilmab as a second-line or above treatment in patients with advanced malignant melanoma and renal cell carcinoma.

To investigate the safety and efficacy of cardunnilizumab in the treatment of advanced mucosal, acral and cutaneous malignant melanoma and advanced renal cell carcinoma.

Primary end point: objective response rate (ORR) Secondary end point: progression-free survival (PFS), disease control rate (DCR), overall survival (OS), incidence of treatment-related adverse events Exploratory study end point: efficacy related marker exploration, gut microbiota or metabolomics changes

ELIGIBILITY:
Inclusion Criteria:

1. Able to sign informed consent;
2. Age ≥18 years, ≤75 years;
3. Cohort 1: histopathologically diagnosed metastatic mucosal or acro-type malignant melanoma with at least second-line prior treatment, including but not limited to PD-1 or PDL1 monoclonal antibody; Cohort 2: histopathologically confirmed metastatic renal cancer with at least second-line prior treatment.
4. There is at least one radiologically measurable lesion according to RECIST1.1 efficacy evaluation criteria;
5. ECOG physical strength score 0-2 points;
6. Expected survival ≥3 months;
7. Major organ function meets the following criteria 7 days before treatment:

   A. Blood routine: neutrophil absolute value ≥1.5×109/L; Hemoglobin ≥80g/L; Platelet ≥90×109/L; B. Blood biochemistry: total bilirubin ≤1.5ULN; ALT and AST≤2.5ULN (Subjects with liver metastases allow ALT or AST≤5×ULN); Serum creatinine ≤1.5ULN or creatinine clearance ≥50ml/min; C. Left ventricular ejection fraction ≥50%; D. Activated partial thromboplastin time (APTT), International Normalized ratio (INR), prothrombin time (PT) ≤1.5ULN; E. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. If baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range may be enrolled F. Myocardial enzyme profiles and troponin within the normal range (simple laboratory abnormalities that are not clinically significant are also allowed to be included)
8. Women of reproductive age should use effective contraception during the study period and for 6 months after the end of the study; A negative serum or urine pregnancy test within 7 days prior to study enrollment; Non-lactating patients; Men should agree to use effective contraception during the study period and for 6 months after the end of the study period;
9. Patients were able to follow the study plan and protocol requirements.

Exclusion Criteria:

1. The presence of symptomatic or untreated known brain metastases or other CNS metastases. Central nervous system metastases that have been shown to be stable or improved after complete resection and/or radiotherapy are not an exclusion criterion, provided that computed tomography (CT) shows stability for at least 4 weeks prior to screening, there is no evidence of cerebral edema and no need for corticosteroids or anticonvulsants;
2. Uncontrolled active infections at the time of screening (such as sepsis, bacteremia, fungemia, viremia, etc.);
3. Active viral hepatitis B or C: Hepatitis B (defined as the presence of hepatitis B core antibody [HBcAb] or hepatitis B surface antigen [HBsAg], and hepatitis B virus DNA [HBV-DNA]) > 1000cps/mL or > lower limit of quantification according to local laboratory methods); Or test positive for hepatitis C (hepatitis C antibodies and/or hepatitis C virus RNA ([RNA]);
4. HIV-infected patients;
5. The patient is known to have systemic vasculitis (e.g., Wegener granuloma, polyarteritis nodosa), systemic lupus erythematosus, co-active or uncontrolled autoimmune disease (e.g., Crohns disease, rheumatoid arthritis, autoimmune hemolytic anemia, etc.), primary or secondary immunodeficiency (e.g., HIV infection or severe symptoms) Infectious diseases, etc.);
6. The patient has a known history of other malignancies;
7. Those who are known to be allergic to the active ingredients or excipients of cardonilizumab in this study;
8. Previously received anti-CTLA-4 specific antibody drug treatment;
9. is currently participating in an interventional clinical study treatment, or has received other investigational drugs or used investigational devices within 4 weeks prior to initial dosing;
10. Received systemic systemic treatment with proprietary Chinese medicines with anticancer indications or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural fluid) within 2 weeks before the first administration;
11. Patients who had systematically used large amounts of glucocorticoids in the 4 weeks prior to enrollment (except those who used inhaled hormones);
12. Serious mental disorders;
13. Patients with serious heart, liver, renal insufficiency, diabetes and other diseases;
14. Pregnant or lactating women;
15. Medical history or evidence of disease that may interfere with the test results, prevent participants from fully participating in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment The investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | From the date of randomization to the date of first documented progression up to 24 months

SECONDARY OUTCOMES:
Progression Free Survival | From the date of randomization to the date of first documented progression up to 24 months
Overall Surviva | From the date of randomization to the date of death from any cause up to 36 months
Disease Control Rate | From the date of randomization to the date of first documented progression up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital, Zhengzhou, China